CLINICAL TRIAL: NCT06284382
Title: Consequence of Early Trauma on Odor Hedonics Appreciation and DOpamine Release
Brief Title: Interaction Between Early Trauma and Odor-induced Dopamine Release
Acronym: T-ODOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022-A02736-37
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, double-blind, parallel-group controlled trial with two arms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presence of early trauma (Other): In the "presence of early trauma" arm, 15 participants are recruited based on a high Childhood Trauma Questionnaire total score.
  Interventions: Other: High score at Childhood Trauma Questionnaire.
- Absence of early trauma (Other): In the "absence of early trauma" arm, 15 participants are recruited based on a low Childhood Trauma Questionnaire total score.
  Interventions: Other: Low score at Childhood Trauma Questionnaire.

INTERVENTIONS:
Other: High score at Childhood Trauma Questionnaire. — In the "presence of early trauma" arm, 15 participants are recruited based on a high Childhood Trauma Questionnaire total score.
  Arms: Presence of early trauma
Other: Low score at Childhood Trauma Questionnaire. — In the "absence of early trauma" arm, 15 participants are recruited based on a low Childhood Trauma Questionnaire total score.
  Arms: Absence of early trauma

SUMMARY:
This prospective, double-blind, parallel-group controlled trial aims to investigate the consequence of early trauma on dopamine release evoked by positive valence odors.

DETAILED DESCRIPTION:
The occurrence of early trauma has been linked to alterations in the development of emotion regulation circuits and functional brain connectivity (particularly in the dorsolateral prefrontal cortex - DLPFC), the dopaminergic response to stress and an alteration in hedonicity (including olfactory hedonicity), which can lead to the onset of psychiatric disorders such as anxiety or depression.

However, few studies have investigated the influence of early trauma on the release of dopamine (DA) evoked by odors with a positive emotional valence. Yet hedonicity is a key component of olfaction, as a positive odor leads to reinforced behavior in areas such as food intake and social interaction. This reinforcement process is thought to be underpinned by the very close link between the olfactory system (olfactory tubercle), the emotional regulation system (DLPFC) and the reward system (striatum), including the release of DA.

The aim of the study is to investigate the influence of early trauma on DAergic transmission evoked by odorants with a positive emotional valence.

To this end, 30 participants will be recruited and divided into two groups: those with early trauma and those without, according to their score on the Childhood Trauma Questionnaire. They will undergo an MRI-PET scan during which they will be exposed to pleasant odors. Subcortical dopaminergic transmission will be analyzed using the PET activity of [11C]Raclopride (a D2 receptor antagonist).

Investigators hypothesize that early trauma resulting in abnormal cortico-subcortical and cortico-cortical connectivity would lead to a deficit in the hedonic appreciation of a pleasant odor, associated with a reduction in DAergic reactivity evoked in the reward system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Have been selected based on the Childhood Trauma Questionnaire score
* Non-smoker
* Be able to speak and read French
* Sign a consent form before intervention.

Exclusion Criteria:

* A pre-existing condition that affects olfaction including congenital anosmia, upper respiratory tract infection, nasal and/or sinus disease,
* Be on medication, with the exception of oral contraceptives
* Pregnant or breast-feeding woman (check with urine pregnancy tests);
* Contraindications to TMS or MRI (implanted medical devices or metallic foreign body in the head);
* Psychiatric disorders
* Use of psychotropic drugs
* Have participated in a study involving the injection of a radiotracer during the year

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Dopamine transmission measured with positron emission tomography | 24 months
  Subcortical dopaminergic transmission will be analyzed, using [11C]raclopride PET activity (D2 receptor antagonist)

SECONDARY OUTCOMES:
Odor hedonic appreciation. | 24 months
  The pleasantness of the odors presented will be assessed on a scale of 1 to 9.
Functional brain connectivity. | 24 months
  Resting-state functional connectivity assessed with fMRI.
Effective brain connectivity | 24 months
  Effective brain connectivity will be assessed using a dual-coil TMS protocol that stimulates the motor cortex and dorsolateral prefrontal cortex during odor presentation. Measurement of the amplitude of the motor response reflects the connectivity between these two regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: JEROME BRUNELIN, Study Director — PSYR2

IPD SHARING:
Plan to Share IPD: No